CLINICAL TRIAL: NCT06802081
Title: TIRO-AF: TIRzepatide for the Treatment of Obesity in Patients With Atrial Fibrillation
Brief Title: TIRzepatide for the Treatment of Obesity in Patients With Atrial Fibrillation
Acronym: TIRO-AF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-228
Record Dates: First submitted 2025-01-27; First posted 2025-01-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Obesity
Keywords: Atrial Fibrillation; Obesity; tirzepatide
MeSH Terms: conditions — Atrial Fibrillation; Obesity | interventions — Tirzepatide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tirzepatide (Experimental): Participants to inject weekly subcutaneous injections of Tirzepatide starting with dose 2.5mg, then increase dose by 2.5mg at week 4 (5mg), week 8 (7.5mg) and at week 12 (10mg) as tolerated.
  Interventions: Drug: Tirzepatide
- Control (Placebo Comparator): Participants to inject weekly subcutaneous injections of normal saline starting with dose 2.5mg, then increase dose by 2.5mg at week 4 (5mg), week 8 (7.5mg) and at week 12 (10mg).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Weekly subcutaneous injections starting with dose 2.5mg, then increase dose by 2.5mg at week 4 (5mg), week 8 (7.5mg) and at week12 (10mg) as tolerated.
  Other Names: Zepbound
  Arms: Tirzepatide
Drug: Placebo — Weekly subcutaneous injections starting with dose 2.5mg, then increase dose by 2.5mg at week 4 (5mg), week 8 (7.5mg) and at week 12 (10mg).
  Other Names: Normal Saline
  Arms: Control

SUMMARY:
This is a single center randomized double blind controlled study of patients (BMI ≥ 27 kg/m2) with obesity and Atrial Fibrillation (AFIB) randomized to Tirzepatide vs. placebo. It is expected that the significant weight loss with Tirzepatide will result in improved control, management, symptom severity, and burden of AFIB at 12 months.

DETAILED DESCRIPTION:
It is estimated that 12 million people in the United States will have AFIB by 2030. The obesity epidemic and all its comorbidities such as hypertension, diabetes and sleep apnea are potent risk factors for AFIB. Weight loss has emerged as a potent treatment for AFIB. This will be a randomized double blind controlled study of patients (BMI≥ 27 kg/m2) with obesity and AFIB randomized to Tirzepatide vs. placebo in the Cleveland Clinic Health System. It is expected that the weight loss with Tirzepatide will result in improved control, management, symptom severity, and burden of AFIB at 12 months.

Patients who met the initial screening criteria (including presence of at least 1% AF burden during a 2 week monitoring period with an ambulatory cardiac monitor) will be invited for possible enrolment. 100 Patients will then be randomized 1:1 to Tirzepatide group versus placebo and will be followed for 12 months. AFIB burden will be assessed through FDA approved event monitor. All patients will receive standard care for management of risk factors as well as nutrition and life style modification counseling.

Management of AFIB including pharmacotherapy, ablation, and direct current cardioversion (DCC) will be at the discretion of Cleveland Clinic's cardiologists.

Patients and investigators will be blinded to treatment assignment. Assessment of the primary endpoint will be based on the blinded downloads and interpretation of event monitors.

The primary objective of the study is to examine Tirzepetide 10mg once a week vs. placebo on severity and symptom burden of AFIB at 12 months.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in this study must meet all of the following criteria:

1. Sinus rhythm at randomization

   1. Sustained normal sinus rhythm (or)
   2. Normal sinus rhythm at office visit
2. Age ≥18 to ≤80 years old
3. BMI ≥ 27 and ≤60 kg/m2
4. AFIB criteria:

   1. Must be documented by ECG or monitor.
   2. Must have symptomatic AFIB (Atrial Fibrillation).
   3. In terms of types of AFIB, either paroxysmal AFIB or persistent AFIB.
5. All anti-diabetic medication (including insulin) must be stable for at least 3 months prior to enrollment,
6. HbA1c ≤10% for patients diagnosed with Type 2 Diabetes Mellitus (T2DM).
7. Ability and willingness to give themselves the medication, comply with study requirements and provide written informed consent.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for inclusion in this study.

1. AFIB ablation within the last 6 months
2. Planned ablation prior to 3 months post randomization
3. Significant cardiac valvular disease with planned cardiac valve intervention/surgery in the next 12 months
4. Severe uncompensated cardiopulmonary disease
5. New York Heart Association Class III or IV
6. Left ventricular ejection fraction <35% at the time of screening
7. Hospitalization in the past 6 months for myocardial infarction, unstable angina, stroke, transient ischemic attack, or heart surgery
8. History of solid organ transplant
9. Type 1 diabetes mellitus or auto-immune diabetes
10. Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m2 at screening or on dialysis
11. Advanced and decompensated cirrhosis characterized by: presence of fibrosis stage 4 (cirrhosis) in liver biopsy, ascites, hepatic encephalopathy, portal hypertension, or esophageal varices.
12. Hemoglobin less than 9 g/dL
13. Current participation or use of investigational therapy or less than 3 months since participation in any drug or device trial.
14. Liver transaminase level >300 U/L
15. Subject reports alcohol use of on average >2 drinks/day
16. Presence of active malignancy (except non-melanoma skin cancer)
17. Life expectancy less than 3 years due to concomitant diseases
18. Major mental health, psychological disorders, or substance abuse disorders that could disqualify the patient from metabolic surgery
19. Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study
20. Plans to move outside the primary location of study (Northeast Ohio) within the next 12 months
21. Any personal or family history of pancreatitis or medullary thyroid cancer or MEN2 (Multiple Endocrine Neoplasia Type 2)
22. Current use or any use within the last 6 months of GLP-1/DPP4i (Glucagon-Like Peptide-1/Dipeptidyl Peptidase-4 inhibitor) or GIP (Gastric Inhibitory Polypeptide)/GLP-1
23. Known hypersensitivity to investigational product due to prior use of GLP-1/DPP4i or GIP/GLP-1
24. Allergy to medical grade tape or adhesive
25. Pregnant, breast-feeding or plans to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
AFib burden | Up to 4 weeks
  Percentage total duration of being in AFIB

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Cho, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No